CLINICAL TRIAL: NCT01997879
Title: An Open-label Study Assessing the Ocular and Systemic Safety and Systemic Absorption of AR-13324 Ophthalmic Solution, 0.02% in Healthy Volunteers
Brief Title: Study Assessing Ocular and Systemic Safety of AR-13324 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AR13324-CS101
Record Dates: First submitted 2013-11-19; First posted 2013-11-28 (Estimated); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AR-13324 Ophthalmic Solution, 0.02% (Experimental): Eyedrop
  Interventions: Drug: AR-13324 Ophthalmic Solution, 0.02%

INTERVENTIONS:
Drug: AR-13324 Ophthalmic Solution, 0.02% — Eyedrop

SUMMARY:
The purpose of this study is to assess systemic safety and absorption of AR-13324 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female subjects at least 18 years of age.
* Within 25% of their ideal weights.
* Medically healthy subjects with clinically insignificant screening results (laboratory profiles, medical histories, ECGs, physical exam) as determined by the Investigator.
* Non-tobacco/nicotine using subjects (minimum of 3 months non-tobacco/nicotine use prior to first dose).
* Subjects with two normal (non-diseased) eyes, defined as nonclinically significant in the opinion of the investigator.
* Intraocular pressure between 14 and 20 mm Hg (inclusive) in each eye at Screening/Qualification.
* Best-corrected visual acuity (BCVA) in each eye of 20/40 or better.
* Willing and able to provide written informed consent prior to any study related procedures and to comply with all study requirements.

Exclusion Criteria:

* Chronic or acute ophthalmic disease including glaucoma, macular degeneration, clinically significant cataract (primary or secondary). Previous cataract surgery.
* Known hypersensitivity to any component of the formulation (benzalkonium chloride, etc.), or to topical anesthetics.
* Previous glaucoma intraocular surgery or glaucoma laser procedures.
* Refractive surgery (e.g., radial keratotomy, PRK, LASIK, etc.).
* Ocular trauma within the past six months, or ocular surgery or laser treatment within the past three months (e.g., laser treatment for glaucoma or retina).
* Evidence of ocular infection, inflammation, cystoid macular edema, clinically significant blepharitis or conjunctivitis at (Screening/ Qualification), or a history of herpes simplex keratitis.
* Ocular medication of any kind within 30 days of Screening/ Qualification
* Any abnormality preventing reliable applanation tonometry of either eye.
* Central corneal thickness greater than 600 µm.
* Cannot demonstrate proper delivery of the eye drop.
* Blood donations or blood loss, within the past 3 months, that would put the patient at risk with the multiple blood samples required in the present study.
* Clinically significant abnormalities in laboratory tests at screening.
* Clinically significant systemic disease (e.g., uncontrolled diabetes, myasthenia gravis, hepatic, renal, cardiovascular or endocrine disorders) which might interfere with the study.
* Participation in any investigational study within the past 30 days prior to screening.
* Changes of systemic medication that could have a substantial effect on IOP within 30 days prior to screening, or anticipated during the study.
* Due to status of preclinical safety program, women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a physician-supervised form of birth control for at least the last two months. An adult woman is considered to be of childbearing potential unless she is one year post-menopausal or three months post-surgical sterilization. All females of childbearing potential must have a negative urine or serum pregnancy test result at the screening examination and must not intend to become pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Assessment | 8 Days
  Blood samples obtained to evaluate the systemic exposure (Area Under the Curve (AUC), Maximum Concentration, Time and half-life (Cmax, tmax and t ½)) to ocularly instilled AR-13324 and its metabolites as appropriate.

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Phoenix, Arizona, United States